CLINICAL TRIAL: NCT03821688
Title: Single Anastomosis Sleeve Jejunal Bypass Compared to One Anastomosis Gastric Bypass and Sleeve Gastrectomy as a Treatment for Morbid Obesity
Brief Title: SAS-J Compared to OAGB and LSG as a Treatment for Morbid Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Alaa Mstafa Hassan Sewefy, Assistant professor, Minia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: fac.med.047
Record Dates: First submitted 2019-01-19; First posted 2019-01-30 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SAS-JB (Experimental): laparoscopic single anastomosis sleeve jejunal bypass
  Interventions: Procedure: SAS-JB
- MGB (Active Comparator): laparoscopic mini gastric bypass
  Interventions: Procedure: OAGB
- LSG (Active Comparator): laparoscopic sleeve gastrectomy
  Interventions: Procedure: LSG

INTERVENTIONS:
Procedure: SAS-JB — single anastomosis sleeve jejunal bypass
  Arms: SAS-JB
Procedure: OAGB — one anastomosis gastric bypass
  Arms: MGB
Procedure: LSG — laproscopic sleeve gastrectomy
  Arms: LSG

SUMMARY:
150 morbidly obese patients divided into to equal groups, group A underwent single anastomosis sleeve jejunal bypass and group B underwent mini gastric bypass, group C underwent sleeve gastrectomy. All patients were followed for at least one year. all cases were evaluated as regard BMI, complications, nutritional status and obesity-related comorbidities.

DETAILED DESCRIPTION:
150 morbidly obese patients divided into to equal groups, group A underwent single anastomosis sleeve jejunal bypass and group B underwent mini gastric bypass, group C underwent sleeve gastrectomy. All patients were followed for at least one year. all cases were evaluated as regard BMI, complications, nutritional status and obesity-related comorbidities. the minimal follow up period is one year

ELIGIBILITY:
Inclusion Criteria:

* obese patients with BMI more than 40 with or without co-morbidity or more than 35 with co-morbidity
* patients fit for laparoscopic surgery
* give approval to share in the study

Exclusion Criteria:

* patients refused to share in the study
* patients unfit for surgery
* patients aged less than 18 and older than 60
* patient with previous upper abdominal surgery either for obesity or other diseases
* revisional bariatric procedures

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
percentage of excess weight loss | 12 months
  percentage of excess weight loss in kilogram

SECONDARY OUTCOMES:
the incidence of nutritional deficiency | 2 years
  the incidence of nutritional deficiency like anemia, hypocalcamia, hypoproteinemia.
the rate of improved co morbidity | 2 years
  the effect of the operation on co morbidity like diabetes and hypertension
the incidence of early operative complications | one month
  early operative complications like leak, bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Alaa M Sewefy, MD, Principal Investigator — Minia University
Locations (1):
- Faculty of medicine, Minya, Egypt